CLINICAL TRIAL: NCT07368855
Title: Changes in Psychiatric Symptoms, Eating Disorder Behaviors, and Health Behaviors Following Six Months of GLP-1 Treatment for Obesity
Brief Title: GLP-1 Medicines and Mental Health Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Thomas Rutledge, Professor in Residence/Staff Psychologist, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E250185
Record Dates: First submitted 2026-01-20; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Depression; GLP-1
Keywords: Veterans, obesity, GLP-1, depression, mental health
MeSH Terms: conditions — Obesity; Depression; Psychological Well-Being | interventions — Glucagon-Like Peptide 1

STUDY DESIGN:
Intervention Model Description: This study consisted of a retrospective observational study of participants receiving GLP-1 medicines for the treatment of obesity. We compared participants to their own baseline (i.e., status at the beginning of their GLP-1 treatment) to evaluate changes in psychiatric and eating disorder symptoms and health-related quality of life after six months of treatment. Participants consisted of US military veterans receiving care from a specialized weight management program in a large Veterans Affairs (VA) hospital in San Diego, California. To be eligible for GLP-1 treatment through the clinic, all veterans had previously completed lifestyle modification education and met national VA pharmacy criteria for having a diagnosis of obesity with one or more weight-related metabolic health conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GLP-1 medicine (Other): GLP-1 treatment
  Interventions: Drug: GLP-1

INTERVENTIONS:
Drug: GLP-1 — Wegovy or Zepbound

SUMMARY:
Key question: Is the use of GLP-1 weight loss medicines - semaglutide and tirzepatide - associated with improvements in mental health and health-related quality of life?

Key finding: Across six- months of GLP-1 treatment, participants reported statistically significant improvements in mental health, eating disorder symptoms, and health-related quality of life domains such as pain interference and sleep quality.

Message for readers: Although GLP-1 medicines are prescribed primarily for weight loss and metabolic health benefits, growing evidence suggests that these medicines may also facilitate meaningful improvements in mental health and quality of life.

DETAILED DESCRIPTION:
In a sample of veterans with obesity and established metabolic disease receiving supervised GLP-1 treatment for weight loss, we observed a consistent pattern of improved psychiatric health, eating disorder behaviors, and health-related quality of life. In addition to observing statistically significant changes across all the latter dimensions using validated psychometric measures, effect size magnitudes were also large enough to suggest potentially clinically meaningful improvements. Importantly, we observed robust evidence of decreases in depressive symptoms - averaging 30% declines in symptom severity - with no signs of increased suicidal ideation symptoms in the sample. The smaller size of this sample necessarily warrants additional research to validate these findings across the broader veteran population and among non-veteran samples.

ELIGIBILITY:
Inclusion Criteria:

* Veterans receiving care at the VA San Diego Healthcare System

Exclusion Criteria:

* VASDHS Veterans not receiving GLP-1 medicines for obesity through the weight control clinic

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory-2 | Six months
  Changes in BDI-2 scores

CONTACTS AND LOCATIONS:
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Data belong to VA San Diego and are not mine to share.